CLINICAL TRIAL: NCT05342545
Title: Electronic Alert-Based Computerized Decision Support to Increase Detection of Chronic Kidney Disease in Patients With Type II Diabetes Mellitus (CKD-DETECT)
Brief Title: Decision Support for Detection of Chronic Kidney Disease in Type II Diabetes Mellitus
Acronym: CKD-DETECT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Brigham and Women's Hospital (Other)
Collaborators: Bayer (Industry)
Responsible Party: Principal Investigator, Gregory Piazza, MD, MS, Associate Director, Thrombosis Research Group, Brigham and Women's Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Diagnostic
Other Study IDs: 2022P000778
Record Dates: First submitted 2022-04-18; First posted 2022-04-22 (Actual); Last update posted 2025-11-04 (Actual); Status verified 2025-11

CONDITIONS: Chronic Kidney Diseases; Type2Diabetes
Keywords: chronic kidney disease; diabetes; urine albumin to creatinine ratio
MeSH Terms: conditions — Renal Insufficiency, Chronic; Diabetes Mellitus

STUDY DESIGN:
Intervention Model Description: 1:1 allocation ratio, randomized controlled trial
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: double-blind
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Alert (Experimental): For patients randomly assigned to the BPA intervention group (alert group), an on-screen electronic alert will be issued during the outpatient clinical encounter that notifies the responsible provider that his or her T2DM patient should be evaluated for CKD with UACR assessment. The provider then will be given on-screen options to either order a UACR assessment or follow a link to learn more about CKD assessment in T2DM. Should the alert-recipient elect to omit an order for UACR assessment and decline to follow a link to learn more about CKD assessment in T2DM, the provider will be able to continue on with clinic visit-related EHR documentation but will need to select an acknowledge reason (rationale) for not following the evidence-based clinical practice recommendation highlighted in the alert.
  Interventions: Other: Alert-based computerized decision support
- No Alert (No Intervention): Providers in the "No Alert" group will not receive any on-screen notification

INTERVENTIONS:
Other: Alert-based computerized decision support — For patients randomly assigned to the BPA intervention group (alert group), an on-screen electronic alert will be issued during the outpatient clinical encounter that notifies the responsible provider that his or her T2DM patient should be evaluated for CKD with UACR assessment. The provider then will be given on-screen options to either order a UACR assessment or follow a link to learn more about CKD assessment in T2DM. Should the alert-recipient elect to omit an order for UACR assessment and decline to follow a link to learn more about CKD assessment in T2DM, the provider will be able to continue on with clinic visit-related EHR documentation but will need to select an acknowledge reason (rationale) for not following the evidence-based clinical practice recommendation highlighted in the alert.
  Other Names: EPIC Best Practice Advisory
  Arms: Alert

SUMMARY:
While data from the National Health and Nutrition Examination Survey (NHANES) estimate that 36.9% of patients with diabetes have CKD, only approximately 10% of patients are aware of their kidney disease. In its 2020 Standards of Medical Care in Diabetes, the ADA recommends that all patients with type II diabetes (T2DM) undergo annual measurement of urine albumin-to-creatinine ratio (UACR). The National Kidney Foundation (NKF) has also proposed an update to the requirements for assessment of adults with diabetes including both an estimated glomerular filtration rate (eGFR) and uACR. The goal of accurately identifying patients with T2DM and CKD is to help providers intervene at an earlier stage of kidney impairment, improve renal outcomes, and reduce associated healthcare costs.

Failure to adopt these guideline recommendations has widespread implications, including underestimation of the burden of CKD in the T2DM population, delays in diagnosis of renal impairment, and ultimately, underutilization of therapies that could improve clinical outcomes. This single-center, 400-patient, randomized controlled trial will assess the impact of an EPIC Best Practice Advisory (BPA; alert-based CDS tool) on guideline-directed assessment for CKD using UACR in patients with T2DM who have not had a UACR in the past year.

DETAILED DESCRIPTION:
The study is a 400-patient single-center Quality Improvement Initiative in the form of a randomized controlled trial of an EPIC EHR BPA. The allocation ratio will be 1:1 for an EPIC BPA versus no notification with randomization by Attending Physician of Record, using odd or even provider ID number, to minimize cluster-effect. While the study will randomize patients by Attending Physician of Record, the observational unit will be the patient.

The study will use a BPA within EPIC that will integrate with the EHR medical history, visit diagnoses, and problem list to identify outpatients with a diagnosis of T2DM and without an established diagnosis of CKD. The BPA will then search the laboratory results section of the EHR for a UACR result within the last year. If the patient with T2DM has not had a UACR result within the past year, he or she will be randomly assigned to the BPA intervention group (alert group) or the control (no alert) group according the Attending Physician of Record's provider ID number. For patients randomly assigned to the BPA intervention group (alert group), an on-screen electronic alert will be issued during the outpatient clinical encounter that notifies the responsible provider that his or her T2DM patient should be evaluated for CKD with UACR. The provider then will be given on-screen options to either order a UACR or follow a link to learn more about CKD assessment in T2DM.

ELIGIBILITY:
Inclusion Criteria:

* BWH outpatients at least 18 years of age who are evaluated in Primary Care or Brigham Medical Specialties Clinics (Cardiovascular Medicine, Endocrinology, and Diabetology) AND
* have a diagnosis of T2DM AND
* have not had a UACR measured in the past year

Exclusion Criteria:

* have an established diagnosis of CKD (medical history, problem list, or visit diagnosis entry in the EHR) OR
* who are undergoing renal replacement therapy (either hemodialysis or peritoneal dialysis) as UACR will be unlikely to result in diagnosis change or therapeutic intervention OR
* who have undergone renal transplantation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400 (Actual)
Dates: Start 2022-12-01 (Actual); Primary Completion 2024-12-31 (Actual); Study Completion 2025-05-30 (Actual)

PRIMARY OUTCOMES:
Frequency of UACR testing order for CKD in patients with T2DM who have not had such testing within the past year | 90 days
  Review the order entry section of the Electronic Health Record (EPIC) to make this determination

SECONDARY OUTCOMES:
Frequency of new clinical diagnosis of CKD in patients with T2DM who have not had UACR assessment within the past year | 90 days
  Review the medical history and problem list sections of the Electronic Health Record (EPIC) to make this determination

OTHER OUTCOMES:
Frequency of prescription of medical therapy for CKD in patients with T2DM, including GLP-1 receptor agonists, renin-angiotensin system antagonists (ACEi or ARB), SGLT2 inhibitors, statins, and emerging anti-inflammatory/anti-fibrotic agents | 90 days
  Review the order entry system for new prescriptions
Frequency of referral to a nephrologist | 90 days
  Review the order entry system for new referrals

CONTACTS AND LOCATIONS:
Locations (1):
- Brigham and Women's Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No